CLINICAL TRIAL: NCT00690820
Title: A Double-blind, Randomized, Multi-center, Placebo-controlled, Cross-over Study to Assess the Efficacy and Safety of Pancrelipase Delayed Release 12,000 Unit Capsules in Subjects Aged 7 - 11 With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Brief Title: Study Investigating a Delayed-Release Pancrelipase in Patients With Pancreatic Exocrine Insufficiency (PEI) Due to Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Djenane Bennett, Solvay Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S245.3.127
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-02

CONDITIONS: Cystic Fibrosis; Pancreatic Exocrine Insufficiency
Keywords: Cystic Fibrosis; Pancreatic Exocrine Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pancrelipase Delayed Release
- B (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Pancrelipase Delayed Release — 12,000 unit Capsules, dosed individually based on fat intake.
  Arms: A
Drug: Placebo Comparator — Placebo
  Arms: B

SUMMARY:
This study will assess the effect of pancrelipase delayed release 12,000 unit capsules on fat and nitrogen absorption in subjects 7 - 11 with pancreatic exocrine insufficiency due to Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CF diagnosis by two positive chloride sweat tests or gene analysis
* Confirmed PEI by historical Coefficient of fat Absorption < 70% without supplementation or current or historical fecal elastase < 50µg/stool (within the last 12 months)
* Currently receiving treatment with a commercially available pancreatic enzyme product on a stable dose for more than 3 months
* Clinically stable condition without evidence of acute respiratory disease or any other acute condition
* Stable body weight and agrees to abstain from sexual activity

Exclusion Criteria:

* Ileus or acute abdomen
* History of fibrosing colonopathy, celiac disease, gastrectomy, Crohn´s disease and small bowel surgery other than minor resection due to meconium ileus without resulting in malabsorption syndrome
* History of distal ileal obstruction syndrome within 6 months of enrollment
* Use of an immunosuppressive drug
* Any type of malignancy involving the digestive tract in the last 5 years
* Known infection with HIV

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (10):
- United States (10):
  - Site 2, Iowa City, Iowa
  - Site 5, Louisville, Kentucky
  - Site 9, Boston, Massachusetts
  - Site 6, Ann Arbor, Michigan
  - Site 4, Minneapolis, Minnesota
  - Site 8, Albuquerque, New Mexico
  - Site 1, Cincinnati, Ohio
  - Site 10, Oklahoma City, Oklahoma
  - Site 7, Oklahoma City, Oklahoma
  - Site 3, Hershey, Pennsylvania

REFERENCES:
- [Result] Graff GR, Maguiness K, McNamara J, Morton R, Boyd D, Beckmann K, Bennett D. Efficacy and tolerability of a new formulation of pancrelipase delayed-release capsules in children aged 7 to 11 years with exocrine pancreatic insufficiency and cystic fibrosis: a multicenter, randomized, double-blind, placebo-controlled, two-period crossover, superiority study. Clin Ther. 2010 Jan;32(1):89-103. doi: 10.1016/j.clinthera.2010.01.012. PMID 20171415
- [Derived] Caras S, Boyd D, Zipfel L, Sander-Struckmeier S. Evaluation of stool collections to measure efficacy of PERT in subjects with exocrine pancreatic insufficiency. J Pediatr Gastroenterol Nutr. 2011 Dec;53(6):634-40. doi: 10.1097/MPG.0b013e3182281c38. PMID 21681115

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in 10 centers in US between June 2008 and October 2008. Before the randomization, subjects were evaluated for eligibility. They underwent a short period of up to 14 days on their usual pancreatic enzyme supplementation.
Pre-assignment Details: Twenty three subjects had given their consent and 17 subjects were randomly allocated to pancrelipase/placebo or placebo/pancrelipase. One subject did not complete the first period of the treatment (consent withdrawal).
Groups:
- Placebo/Pancrelipase: Placebo period followed by Pancrelipase delayed release 12000 units period
- Pancrelipase/Placebo: Pancrelipase delayed release 12000 units period followed by Placebo period
Period: Period 1
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.1) | 8.7 (1.4) | 8.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Fat Absorption (%)
Description: This coefficient is calculated from fat intake and fat excretion : 100*[fat intake-fat excretion]/fat intake. Stools were collected on 3 days during the 5 days treatment period. Higher values indicate a better response.
Time Frame: 5 days
Population: The analysis was done on the Full Analysis Sample defined as the randomized subjects with at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Placebo: Placebo treatment
- Pancrelipase: Pancrelipase delayed release 12000 units treatment
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Percentage | 47.41 (16.84) | 82.81 (8.29)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; The parameter was analyzed using an analysis of variance (ANOVA) including treatment, sequence and period as fixed effect and subject within sequence as a random effect; Test type: Superiority or Other; p < 0.001, ANOVA

2. Secondary Outcome: Coefficient of Nitrogen Absorption (%)
Description: This coefficient is calculated from nitrogen intake and nitrogen excretion : 100*[nitrogen intake-nitrogen excretion]/nitrogen intake. Stools were collected on 3 days during the 5 days treatment period. Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Percentage | 44.98 (20.47) | 80.33 (7.92)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Total Fat Excretion (Grams)
Description: Total amount of fat excreted during the stool collection period. Stools were collected on 3 days during the 5 days treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Grams | 182.9 (68.0) | 58.1 (27.5)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

4. Secondary Outcome: Total Stool Weight (Grams)
Description: Total weight of the stools collected during the stool collection period. Stools were collected on 3 days during the 5 days treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Grams | 436.5 (158.4) | 161.4 (57.5)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Stool Frequency
Description: Stool frequency is the average of the daily number of stools recorded during the treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number per day
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Number per day | 3.46 (1.06) | 1.88 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

6. Secondary Outcome: Percentage of Days With no Flatulence.
Description: The percentage of days with no flatulence is calculated from the diary during the treatment period: 100*(number of days with no flatulence/number of days recorded in diary). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Percentage of days | 36.3 (36.9) | 45.0 (42.1)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.671, ANOVA

7. Secondary Outcome: Percentage of Days With Formed/Normal Stools.
Description: The percentage of days with formed/normal stools is calculated from the diary during the treatment period: 100*(number of days with formed/normal stools/number of days with any stool). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Percentage of days | 38.9 (33.0) | 77.7 (27.0)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, ANOVA

8. Secondary Outcome: Percentage of Days With no Abdominal Pain.
Description: The percentage of days with no abdominal pain is calculated from the diary during the treatment period: 100*(number of days with no abdominal pain / number of days recorded in diary). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 16 | 16
Percentage of days | 65.2 (28.9) | 85.3 (21.1)
Statistical Analysis 1: Comparison: Placebo vs Pancrelipase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, ANOVA

ADVERSE EVENTS:
Time Frame: The adverse events were collected from Screening to the end of the second period of the cross-over trial. A safety follow-up call was performed 5-7 days after the last visit to the clinic.
Description: Only Treatment Emergent Adverse events are presented.
Arm/Group | Placebo | Pancrelipase
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 9/16 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Pancrelipase (N=17)
Rectal Discharge (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Faecal Volume Increased (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Blood glucose increased (Investigations) | 1 | 1
Weight Decrease (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the study to a publisher, reviewer or outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment.